CLINICAL TRIAL: NCT05866367
Title: Measurement of Insulin Levels in Cerebral Spinal Fluid (CSF) of Healthy Adults After a Single Intranasal Dose
Acronym: INI-CSF
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: We are closing this clinical protocol due to supply chain issues. We are no longer able to obtain the intranasal delivery device. We do not have adequate funding available to continue with an alternative intranasal delivery device.
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: A21-299
Record Dates: First submitted 2023-05-05; First posted 2023-05-19 (Actual); Results first posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Healthy
MeSH Terms: interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low dose Intranasal Insulin (Experimental): One dose of 40 international units of regular insulin administered intranasally using the SipNose SP1N1C1 device.
  Interventions: Drug: Low dose Regular Insulin
- High dose Intranasal Insulin (Experimental): One dose of 80 international units of regular insulin administered intranasally using the SipNose SP1N1C1 device.
  Interventions: Drug: High dose Regular insulin

INTERVENTIONS:
Drug: Low dose Regular Insulin — Regular insulin administered intranasally at either 40 IU
  Other Names: Novolin-R
  Arms: Low dose Intranasal Insulin
Drug: High dose Regular insulin — Regular insulin administered intranasally at either 80 IU
  Other Names: Novolin-R
  Arms: High dose Intranasal Insulin

SUMMARY:
The purpose of this study is to find out whether insulin, a drug approved by the FDA for the treatment of diabetes mellitus, reaches the brain and spinal cord when delivered as a nasal spray (intranasally). Intranasal insulin has been shown to improve memory and mood in patients with mild cognitive impairment and dementia, but more evidence is needed to support the ability to effectively target the brain through intranasal routes.

12 healthy adults will be randomly assigned to receive a single dose of either 40 units ("low dose" group) or 80 units ("high dose" group) of insulin. Participants will undergo image-guided lumbar puncture (spinal tap) performed by a study radiologist. Samples of cerebrospinal fluid (a fluid surrounding the brain and spinal cord) and blood will be collected at 5 timepoints during the lumbar puncture: once prior to the administration of intranasal insulin, and again at 10, 20, 30, and 40 minutes after the dose is given. Samples will be tested to determine the level of insulin detected in the cerebrospinal fluid and blood at each time point. Results of this study will provide essential information about the ability of the SipNose device to effectively deliver insulin to the central nervous system of humans as measured in the cerebrospinal fluid.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between ≥18 and ≤ 35 years of age
2. Subject's body mass index is between >=18.5 and <=24.9
3. Subject must be proficient in speaking English to comply with instructions and measures for the study
4. Subject can provide written informed consent
5. Female subjects must have either: (1) a negative pregnancy test at the screening and treatment visits OR (2) be at least 2 years post-menopausal/surgically sterile.

Exclusion Criteria:

1. Subject has medical history and/or clinically determined disorders: chronic sinusitis, previous nasal and/or oto-pharyngeal surgery and severe deviated septum and/or other anomalies.
2. Subject has history of any of the following: active and significant central nervous system, psychiatric illness, pulmonary, or cardiovascular disorders or any other clinically relevant abnormality that inclusion would pose a safety risk to the subject as determined by investigator
3. Subject has participated in a clinical trial investigation within 3 months of this study.
4. Subject has an insulin allergy
5. Subject has Insulin-dependent diabetes
6. Subject is pregnant or breast feeding
7. Contraindication to spinal tap or other safety factors that preclude lumbar puncture in the investigator's opinion

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leah R Hanson, PhD, Principal Investigator — HealthPartners Neuroscience Research
Locations (1):
- HealthPartners Neuroscience Center, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low dose Intranasal Insulin | High dose Intranasal Insulin
Started | 2 | 0
Completed | 2 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study was closed. No high dose individuals were consented prior to closure.
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Intranasal Insulin | High Dose Intranasal Insulin | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex assigned at birth: Male | 0 | 0 | 0
  Sex assigned at birth: Female | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Insulin Concentration Over Time - Cerebrospinal Fluid
Description: Insulin concentration detected in cerebrospinal fluid at 5 time points (pre-insulin dose; and 10, 20, 30 ,40 minutes after dose). Values will be reported as μIU/mL. Higher values indicate a greater concentration of insulin in the cerebrospinal fluid. Concentrations for each time point (overall and by dose) will be reported as a mean +/- standard deviation. The limit of detection of the assay was 0.15mU/L (0.0065µg/L).
Time Frame: 0-40 minutes post-intranasal administration
Population: Study was terminated. No high dose individuals were consented prior to termination.
Measure: Mean (Standard Deviation); unit: µU/ml
Arm/Group | Low dose Intranasal Insulin | High dose Intranasal Insulin
Number analyzed (Participants) | 2 | 0
µU/ml
  0 minutes | 0.57 (0.64) |
  10 minutes | 0.01 (0.01) |
  20 minutes | 0.02 (0.03) |
  30 minutes | 0.05 (0.04) |
  40 minutes | 0 (0) |

2. Primary Outcome: Cmax of Insulin Concentration - Cerebrospinal Fluid
Description: CSF insulin concentration will also be reported by Cmax (peak concentration)
Time Frame: 0-40 minutes post-intranasal administration
Population: Cmax was not summarized as most values were below the limit of detection of the assay.
Measure: Mean (Standard Deviation); unit: uU/mL
Arm/Group | Low dose Intranasal Insulin | High dose Intranasal Insulin
Number analyzed (Participants) | 2 | 0
uU/mL | NA — values below LLOQ |

3. Primary Outcome: Tmax of Insulin Concentration - Cerebrospinal Fluid
Description: CSF insulin concentration will also be reported by Tmax (time of peak concentration)
Time Frame: 0-40 minutes post-intranasal administration
Population: Tmax was not calculated as most values were below the limit of detection of the assay.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Low dose Intranasal Insulin | High dose Intranasal Insulin
Number analyzed (Participants) | 2 | 0
minutes | NA — values below LLOQ |

4. Primary Outcome: AUC (Area Under the Curve) of Insulin Concentration - Cerebrospinal Fluid
Description: CSF insulin concentration will also be reported by AUC (area under the curve, measured as time x concentration).
Time Frame: 0-40 minutes post-intranasal administration
Population: AUC was not calculated as most values were below the limit of detection of the assay.
Measure: Mean (Standard Deviation); unit: uU*min/mL
Arm/Group | Low dose Intranasal Insulin | High dose Intranasal Insulin
Number analyzed (Participants) | 2 | 0
uU*min/mL | NA — values below LLOQ |

5. Secondary Outcome: Insulin Concentration Over Time - Serum
Description: Insulin concentration detected in blood at 5 time points (pre-insulin dose; and 10, 20, 30 ,40 minutes after dose). Values will be reported as μIU/mL. Higher values indicate a greater concentration of insulin in the blood. Concentrations for each time point (overall and by dose) will be reported as a mean +/- standard deviation. Serum insulin concentration will also be reported by Cmax (peak concentration), Tmax (time of peak concentration), and AUC (area under the curve, measured as time x concentration).
Time Frame: 0-40 minutes post-intranasal administration
Population: Study was closed. No high dose individuals were consented prior to closure.
Measure: Mean (Standard Deviation); unit: µU/ml
Arm/Group | Low dose Intranasal Insulin | High dose Intranasal Insulin
Number analyzed (Participants) | 2 | 0
µU/ml
  0 minutes | 5.8 (0.85) |
  10 minute | 10.8 (4.8) |
  20 minutes | 9.75 (3.6) |
  30 minutes | 9.75 (5.16) |
  40 minutes | 9.95 (8.88) |

6. Secondary Outcome: Cmax of Insulin Concentration - Serum
Description: Serum insulin concentration will also be reported by Cmax (peak concentration).
Time Frame: 0-40 minutes post-intranasal administration
Population: Study was closed. No high dose individuals were consented prior to closure.
Measure: Mean (Standard Deviation); unit: uU/ml
Arm/Group | Low dose Intranasal Insulin | High dose Intranasal Insulin
Number analyzed (Participants) | 2 | 0
uU/ml | 10.85 (3.35) |

7. Secondary Outcome: Tmax of Insulin Concentration - Serum
Description: Serum insulin concentration will also be reported by Tmax (time of peak concentration).
Time Frame: 0-40 minutes post-intranasal administration
Population: Study was closed. No high dose individuals were consented prior to closure.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Low dose Intranasal Insulin | High dose Intranasal Insulin
Number analyzed (Participants) | 2 | 0
minutes | 10.0 (0.0) |

8. Secondary Outcome: AUC (Area Under the Curve) of Insulin Concentration - Serum
Description: Serum insulin concentration will also be reported by AUC (area under the curve, measured as time x concentration).
Time Frame: 0-40 minutes post-intranasal administration
Population: Study was closed. No high dose individuals were consented prior to closure.
Measure: Mean (Standard Deviation); unit: uU*min/ml
Arm/Group | Low dose Intranasal Insulin | High dose Intranasal Insulin
Number analyzed (Participants) | 2 | 0
uU*min/ml | 382.25 (115.75) |

ADVERSE EVENTS:
Time Frame: 4 months
Description: Study was terminated. No high dose individuals were consented prior to termination.
Arm/Group | Low dose Intranasal Insulin | High dose Intranasal Insulin
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/0
Other Adverse Events (participants affected / at risk) | 2/2 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low dose Intranasal Insulin (N=2) | High dose Intranasal Insulin (N=0)
Positional Headache (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Headache after lumbar puncture procedure. Required use of blood patch.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low dose Intranasal Insulin (N=2) | High dose Intranasal Insulin (N=0)
Watery eyes (Eye disorders) | 1 (1) | NA
Lightheadedness (Ear and labyrinth disorders) | 2 (2) | NA
Hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | NA
Ear infection (Ear and labyrinth disorders) | 1 (1) | NA
Pain at needle insertion (General disorders) | 1 (2) | NA — after lumbar puncture and after blood patch
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-12): https://cdn.clinicaltrials.gov/large-docs/67/NCT05866367/Prot_SAP_000.pdf